CLINICAL TRIAL: NCT01206517
Title: A Sequential Groups, Open Label, Rising Multiple Dose Study to Assess the Pharmacokinetics, Safety and Tolerability of Sublingual Asenapine in a Pediatric Population With Schizophrenia or Bipolar I Disorder
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Sublingual Asenapine in a Pediatric Population With Schizophrenia or Bipolar I Disorder (P06522 AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06522
Record Dates: First submitted 2010-09-17; First posted 2010-09-22 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: asenapine; pediatric schizophrenia; bipolar I disorder
MeSH Terms: conditions — Schizophrenia | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Participants 10 or 11 years of age
  Interventions: Drug: Asenapine 2.5 mg
- Cohort 2 (Experimental): Participants 10 or 11 years of age
  Interventions: Drug: Asenapine 5 mg
- Cohort 3a-d (Experimental): Cohort 3a: Participants 10 or 11 years of age
  Cohort 3b: Participants 12 or 13 years of age
  Cohort 3c: Participants 14 or 15 years of age
  Cohort 3d: Participants 16 or 17 years of age
  Interventions: Drug: Asenapine 10 mg

INTERVENTIONS:
Drug: Asenapine 2.5 mg — Asenapine tablet, sublingually (SL), 2.5 mg b.i.d. on Days 1-6 and one 2.5 mg tablet, SL, on Day 7.
  Other Names: SCH 900274; Org 5222
  Arms: Cohort 1
Drug: Asenapine 5 mg — Asenapine tablet, SL, 5 mg b.i.d. on Days 1-6 and one 5 mg tablet, SL, on Day 7.
  Other Names: SCH 900274; Org 5222
  Arms: Cohort 2
Drug: Asenapine 10 mg — Asenapine tablets, SL, in a rising dose schedule to 10 mg b.i.d. (with a single 10 mg dose on final day). For Cohorts 3b, 3c and 3d, rising dose schedule begins with asenapine 5 mg b.i.d. on Day 1 and dosing occurs through Day 8. For Cohort 3a, rising dose schedule begins with asenapine 2.5 mg b.i.d. on Day 1 and dosing occurs through Day 12.
  Other Names: SCH 900274; Org 5222
  Arms: Cohort 3a-d

SUMMARY:
This study is an open label, sequential-group, two site, multiple dose escalating study of sublingual administered asenapine in a pediatric population with schizophrenia or bipolar I disorder; in one study cohort (3a) participants with other conditions treatable with chronic antipsychotic medication can also be enrolled. Participants will receive a single sublingual placebo dose on Day -1, followed by multiple sublingual doses of asenapine twice daily (b.i.d.) for 6 days (Cohorts 1 and 2), 7 days (Cohort 3b-d), or 11 days (Cohort 3a), and a final once daily administration on Day 7 (Cohorts 1 and 2), Day 8 (Cohort 3b-d) or Day 12 (Cohort 3a).

ELIGIBILITY:
Inclusion Criteria

For participants in Cohorts 1, 2, 3b, 3c and 3d:

* Diagnosis of schizophrenia or bipolar I disorder
* A schizophrenic participant must have a diagnosis of current schizophrenia of paranoid disorganized, catatonic, or undifferentiated subtype as determined by a structured clinical interview at screening
* A bipolar I disorder participant must have a primary diagnosis of bipolar I disorder, current episode manic, or mixed as determined by a structured clinical interview at screening

For participants in Cohort 3a:

* Documented history of schizophrenia, bipolar disorder, autism, conduct disorder, oppositional defiant disorder, or any condition for which the chronic use of antipsychotic medication (e.g, risperidone, olanzapine, aripiprazole, haloperidol) was warranted and/or administered

All participants:

* Must be at least 10 and not older than 17 years of age at the day of first asenapine dosing (Cohort 3); for Cohort 1 and 2 subjects should be at least 10 and not older than 11 years of age at the day of first asenapine dosing
* Must be able and willing to sign an informed assent as required by local regulations before study participation and able to adhere to dose and visit schedules or their parent/authorized legal representative(s) should be able and willing to sign an informed consent, and should be fluent in the language of the informed consent
* Must have a caregiver or an identified responsible person who is considered reliable by the investigator and who has agreed to provide support to the subject to ensure compliance with trial treatment, outpatient visits, and protocol procedures
* Must be fluent in the language of the investigator, trial staff (including raters) and the informed assent
* Must be willing to discontinue all psychotropic medication during the treatment period except for those specified in the protocol
* Have discontinued the use of strong inhibitors or inducers of cytochrome P450 (CYP)1A2 and/or CYP2D6 (e.g. fluvoxamine, citalopram, fluoxetine, paroxetine, omeprazole, and rifampicin) and beta-blockers, applying a washout period of 5 half lives or 7 days, whichever is longer, AND be stabilized on non-interacting alternative medication (i.e. medication not interacting with asenapine pharmacokinetics) for 2 weeks prior to baseline if their medical condition requires this
* Clinical laboratory tests (complete blood count [CBC], blood chemistry, and urinalysis) must be within normal limits or clinically acceptable to the investigator, after discussion with the Sponsor and following agreement of the Sponsor's medical monitor
* Screening 12 lead electrocardiogram (ECG) conduction intervals and vital signs recordings (oral body temperature, systolic/diastolic blood pressure and pulse rate) must be clinically acceptable according to the investigator, after discussion with the Sponsor and following agreement of the Sponsor's medical monitor
* If male, and non-vasectomized, must agree to use a condom with spermicide (when marketed in the country) or abstain from sexual intercourse, during the trial and for 3 months after stopping the medication

Female participants must:

If unsterilized, have used a medically accepted method of contraception for 3 months (or abstained from sexual intercourse) prior to the screening period, and agree to use a medically accepted method of contraception during the trial (including the screening period prior to receiving trial medication) and for 2 months after stopping the trial medication. An acceptable method of contraception includes one of the following:

* stable oral, transdermal, injectable, or sustained-release vaginal hormonal contraceptive regimen without breakthrough uterine bleeding for 3 months prior to Screening; in addition, during study use of condom and/or spermicide (when marketed in the country)
* intrauterine device (inserted at least 2 months prior to Screening visit); in addition, during study use of condom and/or spermicide (when marketed in the country)

Note: Vasectomy of the partner is not considered sufficient contraception and one of the 2 methods listed above must be used

Females who are not currently sexually active must also consent to use one of these accepted methods of contraception should they become sexually active while participating in the study

* condom (male or female) with spermicide (when marketed within the country),
* diaphragm or cervical cap with spermicide (when marketed within the country) and condom (male),

Exclusion Criteria

The participant will be excluded from entry if ANY of the criteria listed below are met at baseline

The participant:

* Is pregnant, intends to become pregnant (within 3 months of ending the study), or is breastfeeding
* In the opinion of the investigator, will not be able to participate optimally in the study
* Has an uncontrolled, unstable clinically significant medical condition (e.g., renal, endocrine, hepatic, respiratory, cardiovascular, hematologic, immunologic, gastrointestinal or cerebrovascular disease, or malignancy) that may interfere with the interpretation of pharmacokinetic, safety and tolerability evaluations in the opinion of the investigator
* Has a history of any infectious disease within 4 weeks prior to drug administration that in the opinion of the investigator, affects the subject's ability to participate in the trial
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Has a positive screen for drugs with a high potential for abuse (during the Screening period or clinical conduct of the trial)
* Has a history of psychiatric or personality disorders that in the opinion of the investigator and sponsor, affects the subject's ability to participate in the trial
* Has a history of neuroleptic malignant syndrome
* Has a diagnosis of mental retardation or organic brain disorder
* Has a primary diagnosis other than schizophrenia or bipolar I disorder, current episode manic or mixed, that is primarily responsible for current symptoms and functional impairment; this exclusion is not applicable to participants in Cohort 3a
* Has a diagnosis of psychotic disorder or a behavioral disturbance thought to be substance induced or due to substance abuse
* Has a current (past 6 months) substance and alcohol abuse or dependence (excluding nicotine and caffeine)
* Has a history of tardive dyskinesia or tardive dystonia
* If has attention-deficit/hyperactivity disorder (ADHD), has not been on a stable dose of stimulants (e.g. amphetamines, methylphenidate) for the last 3 months (participants who have not taken any stimulants in the last month will not be excluded)
* Has a history of alcohol or drug abuse in the past 2 years
* Has donated blood in the past 60 days
* Has previously received asenapine
* Is at imminent risk of self-harm or harm to others, in the investigator's opinion based on clinical judgment
* Report at Screening, suicidal ideation, or suicidal behavior in the past 6 months
* Is currently participating in another clinical study or have participated in a clinical study (e.g., laboratory or clinical evaluation) within 30 days of baseline
* Is part of the study staff personnel or family members of the study staff personnel
* Has demonstrated allergic reactions (eg, food, drug, atopic reactions or asthmatic episodes) which, in the opinion of the investigator and sponsor, interfere with their ability to participate in the trial
* Smokes more than 10 cigarettes or equivalent tobacco use per day
* Has a history of malignancy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-07-18 (Actual); Primary Completion 2011-08-04 (Actual); Study Completion 2011-08-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine 2.5 mg - Cohort 1: Participants 10 or 11 years of age; administered asenapine 2.5 mg b.i.d on Days 1-6 and a single asenapine 2.5 mg dose in the morning on Day 7
- Asenapine 5 mg - Cohort 2: Participants 10 or 11 years of age; administered asenapine 5 mg b.i.d on Days 1-6 and a single asenapine 5 mg dose in the morning on Day 7
- Asenapine 10 mg - Cohort 3a: Participants 10 or 11 years of age; administered asenapine 2.5 mg b.i.d on Days 1-3, asenapine 2.5 mg in the morning and 5 mg in the evening on Day 4, asenapine 5 mg b.i.d. on Days 5-6, asenapine 5 mg in the morning and 10 mg in the evening on Day 7, asenapine 10 mg b.i.d on Days 8-11, and a single asenapine 10 mg dose in the morning on Day 12
- Asenapine 10 mg - Cohort 3b: Participants 12 or 13 years of age; administered asenapine 5 mg b.i.d on Day 1 (an additional day of 5 mg b.i.d could be allowed), asenapine 10 mg b.i.d on Days 2-7, and a single asenapine 10 mg dose in the morning on Day 8
- Asenapine 10 mg - Cohort 3c: Participants 14 or 15 years of age; administered asenapine 5 mg b.i.d on Day 1 (an additional day of 5 mg b.i.d could be allowed), asenapine 10 mg b.i.d on Days 2-7, and a single asenapine 10 mg dose in the morning on Day 8
- Asenapine 10 mg - Cohort 3d: Participants 16 or 17 years of age; administered asenapine 5 mg b.i.d on Day 1 (an additional day of 5 mg b.i.d could be allowed), asenapine 10 mg b.i.d on Days 2-7, and a single asenapine 10 mg dose in the morning on Day 8
Period: Overall Study
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a | Asenapine 10 mg - Cohort 3b | Asenapine 10 mg - Cohort 3c | Asenapine 10 mg - Cohort 3d
Started | 6 | 6 | 6 | 4 | 4 | 4
Completed | 6 | 6 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a | Asenapine 10 mg - Cohort 3b | Asenapine 10 mg - Cohort 3c | Asenapine 10 mg - Cohort 3d | Total
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 4 | 4 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (0.4) | 10.5 (0.8) | 10.3 (0.5) | 12.5 (0.6) | 14.5 (0.6) | 16.5 (0.6) | 12.1 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 2 | 2 | 2 | 13
  Male | 4 | 3 | 4 | 2 | 2 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Asenapine
Description: Cmax is the peak plasma concentration following a dose of the study drug.
Time Frame: Predose (0 hours) and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 36 and 48 hours after the final asenapine dose (administered on Day 7 for Cohorts 1 and 2; on Day 8 for Cohorts 3b, 3c and 3d; and on Day 12 for Cohort 3a)
Population: All participants administered asenapine with evaluable pharmacokinetic data. Two participants in Cohort 3a and one participant in Cohort 3c did not complete the study and are excluded from pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a | Asenapine 10 mg - Cohort 3b | Asenapine 10 mg - Cohort 3c | Asenapine 10 mg - Cohort 3d
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 3 | 4
ng/mL | 1.84 (1.17) | 3.48 (0.629) | 9.24 (5.17) | 6.75 (0.701) | 6.98 (6.46) | 7.87 (2.68)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Asenapine
Description: tmax is the time from dosing to maximum plasma drug concentration levels.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a | Asenapine 10 mg - Cohort 3b | Asenapine 10 mg - Cohort 3c | Asenapine 10 mg - Cohort 3d
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 3 | 4
hr | 1.0 [0.5 to 2.0] | 1.8 [1.5 to 3.0] | 1.5 [0.5 to 1.5] | 1.0 [1.0 to 1.0] | 0.5 [0.5 to 3.0] | 1.0 [0.5 to 1.5]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 12 Hours Post Dose (AUC0-12) of Asenapine
Description: AUC0-12 is the area under the plasma drug-concentration time curve calculated for the 12 hour interval after dosing.
Time Frame: Predose (0 hours) and 0.5, 1, 1.5, 2, 3, 4, 6 and 12 hours after the final asenapine dose (administered on Day 7 for Cohorts 1 and 2; on Day 8 for Cohorts 3b, 3c and 3d; and on Day 12 for Cohort 3a)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a | Asenapine 10 mg - Cohort 3b | Asenapine 10 mg - Cohort 3c | Asenapine 10 mg - Cohort 3d
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 3 | 4
hr*ng/mL | 11.4 (6.10) | 23.6 (4.02) | 55.2 (20.9) | 41.3 (9.59) | 36.5 (36.7) | 41.8 (12.6)

4. Primary Outcome: Terminal Phase (Elimination) Half-life (t1/2) of Asenapine
Description: Elimination t1/2 is the time it takes for the concentration of the drug in the body to decrease by half during the elimination phase.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a | Asenapine 10 mg - Cohort 3b | Asenapine 10 mg - Cohort 3c | Asenapine 10 mg - Cohort 3d
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 3 | 4
hr | 22.0 (6.12) | 18.5 (3.11) | 15.9 (2.34) | 16.5 (3.38) | 24.3 (14.9) | 24.6 (11.1)

ADVERSE EVENTS:
Time Frame: Up to Day 14
Groups:
- Asenapine 10 mg - Cohort 3a-d: Participants 10-17 years of age:
  Participants 10 or 11 years of age (Cohort 3a); administered asenapine 2.5 mg b.i.d on Days 1-3, asenapine 2.5 mg in the morning and 5 mg in the evening on Day 4, asenapine 5 mg b.i.d. on Days 5-6, asenapine 5 mg in the morning and 10 mg in the evening on Day 7, asenapine 10 mg b.i.d on Days 8-11, and a single asenapine 10 mg dose in the morning on Day 12
  Participants 12-17 years of age (Cohort 3b-d); administered asenapine 5 mg b.i.d on Day 1 (an additional day of 5 mg b.i.d could be allowed), asenapine 10 mg b.i.d on Days 2-7, and a single asenapine 10 mg dose in the morning on Day 8
Arm/Group | Asenapine 2.5 mg - Cohort 1 | Asenapine 5 mg - Cohort 2 | Asenapine 10 mg - Cohort 3a-d
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/18
Other Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 11/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 2.5 mg - Cohort 1 (N=6) | Asenapine 5 mg - Cohort 2 (N=6) | Asenapine 10 mg - Cohort 3a-d (N=18)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 9 (80)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Salivary Hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 7 (8)
Dysgeusia (Nervous system disorders) | 1 (9) | 0 (0) | 7 (37)
Dystonia (Nervous system disorders) | 0 (0) | 4 (5) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 2 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 2 (2) | 2 (2) | 1 (2)
Somnolence (Nervous system disorders) | 1 (4) | 0 (0) | 7 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may not publish/publicly present interim results without prior consent of Sponsor. Any materials that report results of the study must be sent to Sponsor 45 days prior to submission for publication/presentation. Sponsor has right to review and comment. In case of any disagreements concerning appropriateness of the materials, investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues or disagreement, prior to submission for publication/presentation.